CLINICAL TRIAL: NCT05677971
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Fazirsiran in the Treatment of Alpha-1 Antitrypsin Deficiency-Associated Liver Disease With METAVIR Stage F2 to F4 Fibrosis
Brief Title: Study to Check the Safety of Fazirsiran and Learn if Fazirsiran Can Help People With Liver Disease and Scarring (Fibrosis) Due to an Abnormal Version of Alpha-1 Antitrypsin Protein
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-999-3001; 2022-501943-34-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Alpha1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fazirsiran (Experimental): Participants will receive fazirsiran 200 milligram per milliliter (mg/ml) subcutaneous (SC) injection on Day 1, at Week 4, and then every 12 weeks (Q12 W) thereafter up to Week 196.
  Interventions: Drug: Fazirsiran Injection
- Placebo (Placebo Comparator): Participants will receive placebo on Day 1, at Week 4, and Q12 W thereafter up to Week 196.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fazirsiran Injection — Participants will receive fazirsiran 200 mg/ml SC injection on Day 1, at Week 4, and Q12 W thereafter up to Week 196.
  Other Names: TAK-999, ARO-AAT, ADS-001
  Arms: Fazirsiran
Other: Placebo — Participants will receive placebo (sterile normal saline [0.9% NaCl]) SC injection on Day 1, at Week 4, and Q12 W thereafter up to Week 196.
  Other Names: Sodium chloride
  Arms: Placebo

SUMMARY:
The main aim of this study is to learn if fazirsiran reduces liver scarring (fibrosis) compared to placebo. Other aims are to learn if fazirsiran slows down the disease worsening in the liver, to get information on how fazirsiran affects the body (called pharmacodynamics), to learn if fazirsiran reduces other liver injury (inflammation) and the abnormal Z-AAT protein in the liver, to get information on how the body processes fazirsiran (called pharmacokinetics), to test how well fazirsiran works compared with a placebo in improving measures of liver scarring including imaging and liver biomarkers (substances in the blood that the body normally makes and help show if liver function is improving, staying the same, or getting worse) as well as to check for side effects in participants treated with fazirsiran compared with those who received placebo.

Participants will either receive fazirsiran or placebo. Liver biopsies, a way of collecting a small tissue sample from the liver, will be taken twice during this study.

ELIGIBILITY:
Inclusion criteria:

* The participant must have a diagnosis of the Z allele homozygotes (PiZZ) genotype AATD. PiZZ diagnosis from source verifiable medical records is permitted. Otherwise, participants must undergo PiZZ confirmatory testing (genotyping for PiS and PiZ alleles) at screening. PiMZ or PiSZ genotypes are not permitted.
* The participant, of any sex, is aged 18 to 75 years, inclusive.
* The participant's liver biopsy core sample collected should meet the requirements of the protocol.
* The participant has evidence of METAVIR stage F2, F3, or F4 liver fibrosis, evaluated by a centrally read baseline liver biopsy during the screening period; or confirmed as meeting all the entry criteria by central reading of a previous biopsy conducted within 6 months before the estimated enrollment date using an adequate liver biopsy and slides as defined in the study laboratory manual.
* The participant has a pulmonary status meeting the protocol's requirements.
* It must be confirmed that the participant does not have HCC. Participants will be screened for HCC with alpha-fetoprotein (AFP) and abdominal ultrasound. If the participant has any of the following, they will be required to have contrast-enhanced CT or MRI imaging to exclude HCC before randomization.
* An adult participant must have a body mass index (BMI) between 18.0 and 39.0 kilograms per meter square (kg^m2), inclusive.
* The participant is a nonsmoker for at least 6 months before screening.

Exclusion Criteria

* The participant has a history of liver decompensating events (overt hepatic encephalopathy [West Haven Grade >=2] documented by a physician, clinically significant ascites, spontaneous bacterial peritonitis, GI bleeding from varices, hepatopulmonary syndrome, hepatorenal syndrome, portal pulmonary hypertension, or bleeding portal hypertensive gastropathy).
* The participant has a history of the presence of medium or large varices or varices with red wale signs based on a previous esophagogastroduodenoscopy (EGD) within 6 months before the estimated enrollment date. For certain participants, an EGD will be required at screening if there is no EGD available within 6 months before the estimated enrollment date. Presence of small varices with no red wale signs on EGD and no history of bleeding will be acceptable for study eligibility.
* The participant has evidence of other forms of chronic liver diseases, including viral hepatitis B or C, primary biliary cholangitis, primary sclerosing cholangitis, Wilson disease, alcoholic hepatitis, hemochromatosis, liver cancer, history of biliary diversion, or autoimmune hepatitis.
* The participant has alanine transaminase (ALT) or aspartate transaminase (AST) levels >250 units per liter (U/L).
* The participant has a platelet count <60,000 per cubic millimeter (mm^3) (<60 × 10^9 per liter [10^9/L]).
* The participant has albumin <=2.8 gram per deciliter (g/dL) (28 grams per deciliter [g/L]).
* The participant has international normalized ratio (INR) >=1.7.
* The participant is expected to have severe and unavoidable high-level exposure to inhaled pulmonary toxins during the study such as may occur with occupational exposure to mineral dusts or metals.
* The participant has a history of drug abuse (such as cocaine, phencyclidine) within 1 year before the screening visit or has a positive urine drug screen at screening.
* The participant has previously been treated with fazirsiran or any other RNAi for AATD-LD.
* The participant has portal vein thrombosis.
* The participant has a prior transjugular portosystemic shunt procedure.
* The participant has a history of malignancy within the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer. Participants with other curatively treated malignancies who have no evidence of metastatic disease and a greater than 1-year disease-free interval may be entered after approval by the medical monitor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2028-02-17 (Estimated); Study Completion 2030-08-14 (Estimated)

PRIMARY OUTCOMES:
Reduction From Baseline of at Least 1 Stage of Histologic Fibrosis (METAVIR Staging) in the Centrally Read Liver Biopsy at Week 106 in AATD-LD With METAVIR Stage F2 and F3 Fibrosis | Baseline, Week 106
  Reduction from baseline of at least 1 stage of histologic fibrosis METAVIR staging in the centrally read liver biopsy at Week 106 in AATD-LD with METAVIR stage F2 and F3 fibrosis will be assessed.

SECONDARY OUTCOMES:
Percent Change from Baseline in Intrahepatic Z-AAT Protein in Alpha-1 Antitrypsin Deficiency-Associated Liver Disease (AATD-LD) with METAVIR Stage F2 to F3 Fibrosis at Week 106 | Baseline, Week 106
  Percent change from baseline in intrahepatic Z-AAT protein in AATD-LD with METAVIR stage F2 to F3 fibrosis will be assessed.
Reduction From Baseline of at Least 1 Stage of Histologic Fibrosis (METAVIR Staging) in the Centrally Read Liver Biopsy | Baseline, Week 106 and Week 202
  Reduction from baseline of at least 1 stage of histologic fibrosis (METAVIR Staging) in the centrally read liver biopsy in participants with AATD-LD with METAVIR stage fibrosis will be assessed.
Number of Participants With Liver Related Clinical Events up to Week 202 | Baseline up to Week 202
  Number of participants with any qualifying liver-related clinical events up to Week 202 in AATD-LD with METAVIR stage F2 to F4 fibrosis will be assessed.
Change From Baseline in Serum Z-Alpha-1 Antitrypsin (Z-AAT) Protein | Baseline, Week 106, Week 202
  Change from baseline in serum Z-AAT protein in participants with AATD-LD with METAVIR stage fibrosis will be assessed.
Change From Baseline in Intrahepatic Z-AAT Protein Polymer Burden Assessed by Periodic Acid Schiff Plus Diastase (PAS+D) Staining | Baseline, Week 106, Week 202
  Change from baseline in intrahepatic Z-AAT protein polymer burden assessed by PAS+D staining liver biopsy in participants with AATD-LD with METAVIR stage fibrosis will be assessed.
Change From Baseline in Intrahepatic Portal Inflammation | Baseline, Week 106, Week 202
  Change from baseline in intrahepatic portal inflammation liver biopsy in participants with AATD-LD with METAVIR stage fibrosis will be assessed.
Change From Baseline in Vibration-Controlled Transient Elastography (VCTE)/Magnetic Resonance Elastography (MRE)-derived Liver Stiffness | Baseline, Week 106, Week 196 and Week 202
  Change from baseline in VCTE/MRE-derived liver stiffness in participants with AATD-LD with METAVIR stage fibrosis will be assessed.
Change From Baseline in Model of End-Stage Liver Disease (MELD) Score | Baseline, Week 106, and Week 202
  The MELD scoring system is used to assess the severity of chronic liver disease. The MELD score is derived from the participant's serum total bilirubin, serum creatinine, and prothrombin international normalized ratio (INR): 3.78*log e serum bilirubin (milligram per deciliter [mg/dL]) + 11.20* log e INR + 9.57* log e serum creatinine (mg/dL) + 6.43 (constant for liver disease etiology). The MELD score ranges from 6 to 40 with higher scores indicating more severe liver disease and a worse outcome. Change from baseline in MELD score in participants with AATD-LD with METAVIR stage fibrosis will be assessed.
Change From Baseline in Liver Injury | Baseline, Week 106 and Week 202
  Change from baseline in liver injury in participants with AATD-LD with METAVIR stage fibrosis will be assessed.
Percent Change from Baseline in Intrahepatic Z-AAT Protein in AATD-LD With METAVIR Stage F2 to F4 Fibrosis | Baseline, Week 106 and Week 202
  Percent change from baseline in intrahepatic Z-AAT protein in AATD-LD with METAVIR stage F2 to F4 fibrosis will be assessed.
Observed Plasma Concentrations of Fazirsiran | Pre-dose up to Week 220
  Observed Plasma Concentrations of Fazirsiran will be assessed.
Number of Participants with Treatment-emergent adverse event (TEAE) and Serious TEAEs | From start of study drug administration up to end of the study (EOS) (Week 230)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this investigational product (IP) or medicinal product. An SAE is any untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. A TEAE is any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. Number of participants with TEAEs and serious TEAEs will be assessed.
Number of Participants with Clinically Significant Declines in Lung Function Parameters | From start of study drug administration up to EOS (Week 230)
  Standard pulmonary function parameters measured will be used to study lung function.
Change From Baseline in Whole Lung PD15 (15th percentile point) Measured by CT lung Densitometry | Baseline up to Week 196
  Change from baseline in whole lung PD15 (15th percentile point) as measured by CT lung densitometry will be assessed.
Number of Participants with Clinically Significant Change in Vital Signs | From start of study drug administration up to EOS (Week 230)
  Vital signs will include body temperature, respiratory rate, blood pressure, pulse and amount of oxygen in the blood. Any change in vital signs which are deemed clinically significant by the investigator will be reported as AE.
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Parameters | From start of study drug administration up to EOS (Week 230)
  12-lead ECG will be evaluated. Any change in ECG assessments which are deemed clinically significant by the investigator will be reported as AE.
Number of Participants with Clinically Significant Changes in Clinical Laboratory Assessments | From start of study drug administration up to EOS (Week 230)
  Clinical laboratory assessments include hematology, serum chemistry, coagulation, and urinalysis. Changes in laboratory values may be considered as AE if they were judged to be clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (84):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona Thomas D. Boyer Liver Institute, Tucson, Arizona
  - Gastroenterology & Liver Institute, Escondido, California
  - University of California San Diego, Altman Clinical and Translational Institute, La Jolla, California
  - UCLA Pulmonary and Critical Care, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California Benioff Children's Hospital, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Indiana University School of Medicine - Indianapolis, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Morgan Stanley Childrens Hospital of New York Presbyterian (CHONY) - PIN, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texoma Liver Center, Denison, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - VCU Medical Center North Hospital, Richmond, Virginia
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincents Hospital Melbourne - PPDS, Fitzroy, Victoria
- Austria (4):
  - LKH-Universitätsklinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Klinikum Klagenfurt Am Wörthersee, Klagenfurt
  - Medizinische Universität Wien (Medical University of Vienna), Vienna
- Belgium (2):
  - UZ Antwerpen, Antwerp
  - UZ Leuven, Leuven
- Brazil (2):
  - Hospital Sirio-Libanes, São Paulo
  - Universidade Estadual Paulista Julio de Mesquita Filho Faculdade de Medicina Campus de Botucatu, São Paulo
- Canada (3):
  - GI Research Institute, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Inspiration Research Limited, Toronto, Ontario
- Institut klinicke a experimentalni mediciny, Prague, Czechia
- Hvidovre Hospital, Hvidovre, Denmark
- France (6):
  - Hôpital Beaujon, Clichy
  - Hôpital de La Croix Rousse, Lyon
  - Centre Francois Magendie, Pessac
  - Hopital PONTCHAILLOU CHU de Rennes, Rennes
  - Hospital Purpan, Toulouse
  - Hôpital Paul Brousse, Val-de-Marne
- Germany (5):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Charité - Campus Virchow-Klinikum-Ostring 1, Berlin
  - Hannover Medical School, Hanover
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Universitätsklinikum Tübingen, Tübingen
- Beaumont Hospital, Dublin, Ireland
- Italy (3):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Netherlands (2):
  - Amsterdam UMC - VUmc - De Boelelaan, Amsterdam
  - Leiden University Medical Center, Leiden
- Poland (2):
  - ID Clinic Arkadiusz Pisula, Śląskie
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
- Portugal (3):
  - CCA Hospital Braga, Braga
  - Hospital Nélio Mendonça, Funchal
  - Centro Hospitalar do Porto, Porto
- Spain (4):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- Sweden (2):
  - Karolinska Universitetssjukhuset Huddinge, Huddinge
  - Universitetssjukhuset i Linköping, Linköping
- Inselspital Bern, Bern, Switzerland
- United Kingdom (5):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Free Hospital, London
  - King's College Hospital, London
  - Queen's Medical Centre, Nottingham
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/e37eea10ca934732?idFilter=%5B%22TAK-999-3001%22%5D